CLINICAL TRIAL: NCT00725023
Title: A Randomized Double-blind Study to Assess the Use of TDP© Heat-lamp as an Effective Therapy for Tennis Elbow Pain (Lateral Epicondylitis Pain)
Brief Title: Use of TPD Heat Lamp for Tennis Elbow Pain - a Randomized-controlled Trial
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Jyoti Kotecha, Assistand Director, Queen's University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CAM01
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Lateral Epicondylitis
Keywords: Pain, chronic pain, tennis elbow, lateral epicondylitis
MeSH Terms: conditions — Tennis Elbow; Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Treatment: TDP© Lamp used Duration of each treatment 30min Course of treatment 3 times a week for 3-4 weeks
  Interventions: Device: TDP© Lamp
- 2 (Other): Treatment: Dummy TDP© Lamp used Duration of each treatment 30min Course of treatment 3 times a week for 3-4 weeks
  Interventions: Device: Dummy TDP© Lamp

INTERVENTIONS:
Device: TDP© Lamp — TDP© heat lamp is an electrical device with a heating element sitting behind a ceramic plate made of clay and minerals
  Arms: 1
Device: Dummy TDP© Lamp — The dummy TDP© heat lamp is an electrical device with the heating element removed.
  Arms: 2

SUMMARY:
Tennis elbow (Lateral epicondylitis) is a common condition seen in Family Medicine that gives rise to pain, and can lead to loss of function and time off work.

The normal treatment for tennis elbow pain is oral pain relief medication (analgesia), and/or physiotherapy, local massage or even surgery. In mainland China, tennis elbow pain has also been treated using TDP © Heat-lamp therapy, and is considered to be an effective treatment for this condition.

This study is a clinical trial that seeks to measure the effectiveness of the TDP © Heat-lamp therapy to relieve tennis elbow pain without the use of oral pain medication.

DETAILED DESCRIPTION:
Double-blind randomized controlled trial

Patient recruitment

Patients registered in the Electronic Medical Record (EMR) system of the Family Medicine Centre of Queen's University with a confirmed diagnosis of tennis elbow (lateral epicondylitis) in the 12-month period from 1st March 2008 to 31st March 2009, are recruited and studied. An internal email plus paper memo will be circulated to all other Family Physicians in the Centre, requesting their participation in the study. Patients are then selected randomly from the pool.

Entry/Randomization Procedure

All eligible patients enrolled in the study centre will be entered into a patient registration log. This will automatically provide a serial number for that patient that should be used for all documentation and correspondence about this patient. All randomizations will be done centrally by the administrator at the CSPC.

Randomization

A total of 116 patients will be randomized into two equal arms of 58 patients in each. Arm 1 is the trial arm and Arm 2 is the control arm.

Treatment

Arm 1: Patients will be given a four-week course of TDP© Heat-lamp. The heat-lamp will be targeted to the pain site on the elbow. Each treatment will take about 30 minutes.

Arm 2: Patients will be given a four-week course of TDP© Heat-lamp using a dummy TDP© Heat-lamp. A dummy heat-lamp is a modified version of the TDP© Heat-lamp without the intended therapeutic effects. The dummy heat-lamp will be targeted to the pain site on the elbow. Each treatment will take about 30 minutes.

Allocation of Treatment

Treatment is executed by staff nurses at the Centre. The staff nurse will be blinded to the coding of the TDP© Heat-lamps, and will operate the lamp for 30 minutes at a specified distance of 20cm from the surface of the affected limb of each patient.

During the course of treatment, patients will be advised not to use any other means of analgesia. If they do, it must be recorded in a patient diary provided to them for use during the study. Patients that have taken oral medication may be considered to be inadmissible subjects during the final analysis.

Dose Adjustment

There is no dose adjustment permitted. During the treatment, patients will be regularly monitored for the development of any undue discomfort. If discomfort is experienced by a patient, treatment will be terminated immediately.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have consented.
* Patients diagnosed with tennis elbow pain. Definition of tennis elbow (lateral epicondylitis) is "pain or tenderness on loading relevant muscle on the lateral epicondyle, with no shoulder or wrist pain.". Patients recruited will be interviewed and examined to confirm the clinical diagnosis. The level of pain will be assessed with the visual analogue scale (VAS) and level of functional disability with the QUICKDASH Questionnaire.
* Patients must be between the ages of 18-65.

Exclusion Criteria:

* Patients with existing diagnosis of neuropathic pain, metabolic or metastatic bone pain will be excluded. So will patients with recent or previous bone fracture of the elbow and epicondyles.
* Patients taking any form of oral analgesia in the last 2 weeks prior to randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2008-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To determine if TDP© heat lamp is an effective therapy for the alleviation of chronic pain due to lateral epicondylitis (tennis-elbow pain.) | At completion of trial

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Leung, MD, Principal Investigator — Queen's University
Locations (1):
- Queen's University-CPC, 220 Bagot Street, Kingston, Ontario, Canada